CLINICAL TRIAL: NCT05817955
Title: Clinical Study of Azacitidine Combined With Ruxolitinib in the Treatment of Higher-risk Myelodysplastic Syndromes∕Myeloproliferative Neoplasms
Brief Title: Clinical Study of Azacitidine Combined With Ruxolitinib in the Treatment of Higher-risk MDS/MPN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangbin Hospital Affiliated to Jiangsu University (Unknown); Nanjing Second Hospital (Unknown); Jiangning Hospital Affiliated to Nanjing Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-757
Record Dates: First submitted 2023-03-02; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: MDS/MPN
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine (AZA) with Ruxolitinib (Experimental): The treatment phase of each course of treatment is based on Azacitidine (AZA)+Ruxolitinib. Specific scheme: (1) Azacitidine+Ruxolitinib scheme: Azacitidine (AZA) 75mg · m-2 · D-1, D1 to D7, subcutaneous injection; Ruxolitinib, D1 to D28, orally, select Ruxolitinib initial dose according to platelet level: ① PLT> 100X10*9/L: 20mg BID orally; ② PLT (50-100) X10*9/L: 15mg BID orally; ③ PLT <50X10*9/L: 10mg Bid orally.
  The above schemes are all 28 days of treatment. If the patient has serious adverse reactions (such as infection and bone marrow suppression), appropriately delay the next course of treatment or adjust the amount of RUXOLITINIB. Termination of the scheme treatment.
  Interventions: Drug: Azacitidine (AZA) with Ruxolitinib

INTERVENTIONS:
Drug: Azacitidine (AZA) with Ruxolitinib — 1. Antibiotics: Antibiotic treatment is positively given when symptoms related to infection, and other support treatment is strengthened.
  2. Blood products: Infuse the blood products according to the patient's blood routine test. Drugs that need to be used by other diseases must be recorded in detail in the case report form, including the general name of the drug, the dosage of the medication, and the frequency of administration. Drugs are not allowed to be combined: Avoiding the use of granulocyte colony-stimulating factor (G-CSF), there may be risk of spleen rupture.

SUMMARY:
This study observes the safety and efficacy of Azacitidine (AZA) combined with ruxolitinib to treat higher-risk Myelodysplastic Syndromes∕Myeloproliferative Neoplasms(MDS/MPN)

DETAILED DESCRIPTION:
This is an open label, a multi -centered clinical trial, aiming to evaluate the safety and efficacy of Azacitidine with Ruxolitinib to treat MDS/MPN patients Myelodysplastic Syndromes/Myeloproliferative Neoplasms（MDS/MPN） are a set of malignant clonal diseases that originated from hematopoietic stem cells, which have both the characteristics of MDS and MPN. They also have the risk of transforming to Acute Myeloid Leukemia (AML). According to the 2016 World Health Organization (WHO) classification, MDS/MPN include Chronic myelomonocytic leukemia(CMML), Atypical chronic myeloid leukemia(aCML)，Juvenile myelomonocytic leukemia (JMML), MDS/MPN with ring sideroblasts and thrombocytosis(MDS/MPN-RS-T), and MDS/MPN unclassified(MDS/MPN-U). Except for JMML, other types of MDS/MPN mainly happened in persons over 60 years old, and the heterogeneity of the disease is large. At present, the treatment is limited. Although allo hematopoietic stem cell transplantation is the only way to cure the diseases, a recent large series study on CMML showed that allo hematopoietic stem cell transplantation would increase the mortality risk of lower-risk CMML, and did not obtain survival benefit in higher-risk CMML. Therefore, it is currently urgent to explore the new treatment for MDS/MPN.

CMML is the most common subtype of MDS/MPN, manifested the increased monocytes in peripheral blood (absolute cell count ≥1x109/L and percentage ≥10%, which lasts more than 3 months) accompanied with at least one lineage dysplasia and bone marrow blasts ≤20%. The median diagnosis age is (73-75) years old, and the estimated annual incidence in the population is 4/10,000.

The treatment strategy of CMML based on the prognostic stratification. According to the prognostic stratification, low-risk patients (low and inter-1) receive red blood cells transfusion and cytoreductive treatment. For high-risk (inter-2 and high) patients who are unsuitable for stem cell transplantation, hypomethylating agents and clinical trials are recommended. The hypomethylating agents (including Decitabine, Azacitidine, and oral Decitabine) are the only drugs approved by the FDA in the United States for CMML treatment. The approvement were based on MDS clinical trials that included CMML, such as CALGB Studies (including 14 patients with CMML) and European AZA-001 Studies (including 11patients with CMML). Since then, many prospective and retrospective studies containing CMML have confirmed its efficacy. The Overall Response Rates (ORR) is 40-50% for hypomethylating agents, while Complete Remission (CR) is less than 20%. In addition, a recent prospective clinical trial pointed out that hypomethylating agents did not achieved clinical response in MPN-CMML, and no significant difference was found between hypomethylating agents group and Hydroxyurea group in Overall Survivals (OS) and Leukemia Free Survival.

In addition to hypomethylating agents, clinical trials are also recommended for patients with higher risks CMML. At present, several clinical trials including Lenzilumab (GM-CSF monoclonal antibody, NCT02546284), Tipifarnib (Fennec metastases inhibitor, NCT02807272), Ruxolitinib (JAK1/2 inhibitors, NCT03722407) and Cobimetinib (MEK inhibitor, NCT04409639) are carried on in CMML. The results show that they have good efficacy and safety in CMML. In addition, a series of clinical trials combined hypomethylating agents with other drugs to explore the way to increase the efficacy in CMML.

Some MDS/MPN patients have the clinical manifestations of MPNs such as increased blood cells, large spleen sizes, and constitutional symptom. Meanwhile, activated inflammatory cytokine secretion also exists in MDS/MPN. Ruxolitinib is JAK1/JAK2 inhibitor used for the treatment of myelofibrosis. A multi -center phase I clinical trial of ruxolitinib including 20 CMML patients showed that 4 patients obtained hematopoietic improvement, and 1 patient obtained bone marrow PR. Of the 9 patients with splenomegaly, 5 patients received spleen reduction > 50%. 10 of 11 patients with constitutional symptom were significantly improved. The ORR was 35% combining spleen response and MDS/MPN International Working Group (IWG) efficacy criteria. Only one patient had level 3 platelet decrease, indicating that ruxolitinib had less impact on platelet counts in CMML. Based on this, the phase I/II clinical trial was included 50 patients with CMML. The ORR according to MDS/MPN IWG was 38%, and 43% patients achieved spleen reduction. The most common adverse events were anemia (10%) and platelet decrease (6%), further confirming the safety and efficacy of ruxolitinib in the treatment of CMML.

In addition, a phase II clinical trial explores the efficacy of ruxolitinib in aCML (n = 23) and chronic neutrophilic leukemia (CNL) (n = 22). The ORR was 35% (11 PR[9 CNL and 2 aCML], 4 CR [CNL]). The most common 3/4 adverse event was anemia (34%) and platelet decrease (14%). It is worth noting that the efficacy was better in CNL compared with aCML.

Based on previous studies, we intend to further investigate the safety and efficacy of azacitidine combined with ruxolitinib in the treatment of higher-risk myelodysplastic syndromes/myelodysplastic diseases (MDS/MPN).

ELIGIBILITY:
Inclusion Criteria:

• According to WHO (2016) classification, researchers made the diagnosis of CMML based on clinical and morphological characteristics. Other criteria should be met: 1) Neut ≥2x109/L, PLT ≥25x109/L, 2) belongs to the following prognostic risk group according to CPSS-MOL or MMM : CPSS-MOL: inter-2 risk (2 to 3 points); high risk (≥4 points);

MMM: inter-2 risk (2.5 to 4.5 points); high risk (≥5 points), or:

* According to the WHO (2016) classification standards (Arber 2016), researchers made the diagnosis of other types of MDS/MPN (including aCML and MDS /MPN-U) based on clinical and morphological characteristics. Other criteria should be met: 1) Neut ≥2x109/L, PLT ≥25x109/L, 2) Bone marrow blasts ≥5%;
* Patients who are not suitable for hematopoietic stem cell transplantation (HSCT) according to the local medical standards and treatment guidelines;
* Patients who are suitable for Azacitidine(AZA) treatment according to the local medical standards and treatment guidelines;
* BCR-ABL positive Chronic Myelogenous Leukemia (CML) and Ph chromosomal negative classic myeloproliferative Neoplasms, such as essential thrombocytosis (ET), polycythemia vera (PV) and primary myelofibrosis (PMF) are excluded;
* Age is between 18 to 80 years old;
* ALT, AST and serum bilirubin is no more than 2 times of the upper limit of normal values (ULN), serum creatinine is no more than 150 μmol/L, and serum myocardial enzyme is less than (the same age) 2 times of normal value upper limit;
* The LVEF determined by the echocardiography is no less than 50%;
* Estimated glomerular filtration rate (EGFR) is no less than 30ml · min · 1.73m2;
* Eastern Tumor Collaboration Group (ECOG) physical states score is 0 to 2;
* Informed Consent Form is signed by patients or legal agents.

Exclusion Criteria:

* BCR-ABL positive Chronic Myelogenous Leukemia (CML) and Ph chromosomal negative classic myeloproliferative Neoplasms, such as essential thrombocytosis (ET), polycythemia vera (PV) and primary myelofibrosis (PMF) ;
* Low risk or inter-1 risk CMML patients according to CPSS-MOL or MMM scores; other types of MDS/MPN with less than 5% bone marrow blasts;
* Patients with Neut<2x109/L, PLT<25x109/L;
* Secondary acute leukemia, myeloid sarcoma, and blast phase of aCML;
* Patients who are allergic to any drug involved in the trial;
* Pregnancy, lactating Women, and patients who are unwilling to use contraceptives;
* Patients with abnormal Liver and kidney function which exceeded the inclusion criteria;
* Patients with organic heart disease with clinical symptoms or heart dysfunction (NYHA ≥ level 2);
* Patients with other malignancies at the same time except the following situations:

Patients had received treatment for the purpose of cure and had no active malignancies for at least 5 years prior to enrollment; 2)Patients had received sufficient treatment, non-melanoma skin cancer or malignant freckles -like moles with no signs of illness (even if random grouping is less than 3 years); 3)Received sufficient treatment, in situ cancer without signs of illness (even if the random group is less than 3 years);

* Patients with AIDS, syphilis, active hepatitis B (HBV-DNA can be measured) and hepatitis C;
* Patients with cardiovascular diseases with clinical significance, such as arrhythmia that have not been controlled or have symptoms, congestive heart failure or myocardial infarction within 6 months, or level 3 (moderate) or level 4 (Severe) heart disease (NYHA according to the New York Heart Society's functional grading method);
* Patients with any situations that might interfere with research procedures or results, or have the medical status or disease that will bring a certain risk to participating in this study judged by researchers (such as activity systemic infection);
* Patients who can't understand or follow the research plan;
* Patients who are under 18 or over 80 years old;
* Patients who underwent a major surgery within 4 weeks before the random grouping;
* Patients who are participating in other clinical trials one month before joining the group;
* Patients who rely on illegal drugs;
* Patients with psychological disorders or cognitive disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | From randomization to the end of Cycle 6 (each cycle is 28 days)
  Complete remission was achieved according to the remission criteria of MDS/MPN
overall survival | From the time of randomization to time for up to 2 years
  It is measured from the date of randomization to the date of death from any cause; patients not known to have died at least follow-up are censored on the date they were last known to be alive.
overall response rate | From randomization to the end of Cycle 6 (each cycle is 28 days)
  overall response includes all the response according to the remission criteria of MDS/MPN

SECONDARY OUTCOMES:
progression-free survival | From the time of randomization to time for up to 2 years
  The progression-free survival was calculated as the time from randomization to disease recurrence or death due to disease progression
Early mortality | up to 3 months
  Early mortality was defined as death within the first 3 months after initiation of induction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxun Shi, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No